CLINICAL TRIAL: NCT02637999
Title: Randomized Open-label Substudy of Daily Myrcludex B Plus Pegylated Interferon-alpha-2a in Patients With HBeAg Negative Chronic Hepatitis B Co-infected With Hepatitis Delta
Brief Title: Myrcludex B Plus Pegylated Interferon-alpha-2a in Patients With HBeAg Negative HBV/HDV Co-infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hepatera Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYR 201 (HDV)
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Chronic Hepatitis D Infection
MeSH Terms: interventions — peginterferon alfa-2a; myrcludex-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MXB then PEG IFN (Experimental): Myrcludex B 2mg daily for 24 weeks, followed by PEG IFN alfa-2a 180 µg/0.5 mL weekly for 48 weeks
  Interventions: Drug: PEG IFN alfa-2a; Drug: Myrcludex B
- MXB + PEG IFN then PEG IFN (Experimental): Myrcludex B 2mg daily and PEG IFN alfa-2a 180 µg/0.5 mL weekly for 24 weeks, followed by PEG IFN alfa-2a 180 µg/0.5 mL weekly for 24 weeks
  Interventions: Drug: PEG IFN alfa-2a; Drug: Myrcludex B
- PEG IFN (Active Comparator): PEG IFN alfa-2a 180 µg/0.5 mL once weekly for 48 weeks
  Interventions: Drug: PEG IFN alfa-2a

INTERVENTIONS:
Drug: PEG IFN alfa-2a
  Other Names: Pegasys
Drug: Myrcludex B
  Other Names: Myrcludex
  Arms: MXB + PEG IFN then PEG IFN; MXB then PEG IFN

SUMMARY:
Randomized open-label substudy of daily Myrcludex B (MXB) plus pegylated interferon-alpha-2a (PEG-INF-a) in patients with hepatitis B e antigen (HBeAg) negative chronic hepatitis B virus (HBV) co-infected with hepatitis delta virus (HDV).

DETAILED DESCRIPTION:
The study is designed to evaluate safety and efficacy of MXB in a subset of HBV infected patients who are co-infected with HDV. Hepatitis delta represents the most severe form of chronic viral hepatitis and there is no approved treatment option available for patients infected with both HBV and HDV.

24 patients will be randomised into 3 arms: pre-treatment with MXB followed by PEG-INF-a treatment versus a combination of both drugs versus PEG-INF-a.

Prolonged blockade of HBV entry into hepatocytes should also block infection with HDV particles (which uses hepatitis B surface antigen (HBsAg) as its envelope) and thus provide a therapeutic option for this otherwise hardly treatable disease. PEG-INF-a is used for the treatment of chronic hepatitis delta. The study endpoints are virological response (HBsAg, hepatitis delta virus ribonucleic acid (HDV RNA), hepatitis B virus deoxyribonucleic acid (HBV DNA)), as well as safety and tolerability and drug immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B defined by the presence of HBsAg for at least 6 months prior to screening period. Co-infection with hepatitis D virus defined as positive anti-HDV antibodies for at least 3 months and positive for HDV-RNA within the screening period.
* Liver biopsy performed within one year prior to screening or during screening period.
* HBeAg negative
* All women of childbearing potential must have a negative urine pregnancy test prior to enrolment.
* Women must:

  1. Be menopausal for at least 2 years, or
  2. Be surgically sterile (total hysterectomy or bilateral ovariectomy or bilateral tubal ligation/clips or otherwise be incapable of pregnancy), or
  3. Not be heterosexually active during the study, or
  4. Agree to use a highly effective method of birth control (double barrier method or combination of barrier method with hormonal or intrauterine device) during the study and for 3 month after the last dosing of the investigational medicinal product.
* Men must agree to use a highly effective method of birth control (double barrier methods or combination of barrier method with hormonal or intrauterine device in their women-partner) and not to donate a sperm during the study and for 3 month after the last dosing of the investigational medicinal product.
* An understanding, ability and willingness to fully comply with study procedures and restrictions.
* An ability to provide the written informed consent to participate in the study

Exclusion Criteria:

* Decompensated liver disease (Child-Pugh-Score >6).
* Co-infected with hepatitis C virus (HCV), or HIV.
* Patients with presence of anti-HCV antibody and negative HCV RNA in two separate occasions within 12 months prior to screening could be enrolled into the study after sponsor written permission.
* ALT > 6 ULN.
* Creatinine clearance < 60 mL/min.
* Total bilirubin > 2 mg/dL.
* Confirmed contraindication for treatment with PEG-INF-a.
* History of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC, such as suspicious foci on imaging studies or elevated serum alpha-fetoprotein (AFP) levels. In patients with such findings, HCC will be ruled-out prior to screening for the present study.
* One or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, e.g. congestive heart failure or other severe cardiopulmonary disease). Patients with Gilbert's syndrome and Dubin-Johnson syndrome, two benign disorders associated with low-grade hyperbilirubinemia can be enrolled into the trial.
* History of clinically evident pancreatitis.
* History of alcohol or drug abuse within the preceding two years. For the purposes of the present study, alcohol abuse is arbitrarily defined as frequent consumption of alcoholic beverages with an average daily intake of more than 40 g of ethanol.
* Participation in another study with an investigational drug within less than one month prior to this study or simultaneously to this study.
* Patients who are unable or unwilling to follow the protocol requirements.
* Patients with a history of seizures, central nervous system disorders or psychiatric disability thought to be clinically significant in the opinion of the investigator.
* Patients with limited mental capacity to the extent that she/he cannot provide informed consent or information regarding adverse events of the study drug.
* Clinically significant renal, respiratory or cardiovascular disease.
* Pregnancy and lactation.
* Patients who have previously participated in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2016-01-21 (Actual); Study Completion 2016-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Bogomolov, PhD, Principal Investigator — LLC "Clinical Hospital of Tsentrosoyuz"

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavanchy D. Hepatitis B virus epidemiology, disease burden, treatment, and current and emerging prevention and control measures. J Viral Hepat. 2004 Mar;11(2):97-107. doi: 10.1046/j.1365-2893.2003.00487.x. PMID 14996343
- [Background] Yan H, Zhong G, Xu G, He W, Jing Z, Gao Z, Huang Y, Qi Y, Peng B, Wang H, Fu L, Song M, Chen P, Gao W, Ren B, Sun Y, Cai T, Feng X, Sui J, Li W. Sodium taurocholate cotransporting polypeptide is a functional receptor for human hepatitis B and D virus. Elife. 2012 Nov 13;1:e00049. doi: 10.7554/eLife.00049. PMID 23150796
- [Background] Trauner M, Boyer JL. Bile salt transporters: molecular characterization, function, and regulation. Physiol Rev. 2003 Apr;83(2):633-71. doi: 10.1152/physrev.00027.2002. PMID 12663868
- [Background] Romeo R, Del Ninno E, Rumi M, Russo A, Sangiovanni A, de Franchis R, Ronchi G, Colombo M. A 28-year study of the course of hepatitis Delta infection: a risk factor for cirrhosis and hepatocellular carcinoma. Gastroenterology. 2009 May;136(5):1629-38. doi: 10.1053/j.gastro.2009.01.052. Epub 2009 Jan 29. PMID 19208358
- [Background] Cornberg M, Protzer U, Dollinger MM, Petersen J, Wedemeyer H, Berg T, Jilg W, Erhardt A, Wirth S, Schirmacher P, Fleig WE, Manns MP. Prophylaxis, diagnosis and therapy of hepatitis B virus (HBV) infection: the German guidelines for the management of HBV infection. Z Gastroenterol. 2007 Dec;45(12):1281-328. doi: 10.1055/s-2007-963714. No abstract available. PMID 18080231
- [Background] Blank A, Markert C, Hohmann N, Carls A, Mikus G, Lehr T, Alexandrov A, Haag M, Schwab M, Urban S, Haefeli WE. First-in-human application of the novel hepatitis B and hepatitis D virus entry inhibitor myrcludex B. J Hepatol. 2016 Sep;65(3):483-9. doi: 10.1016/j.jhep.2016.04.013. Epub 2016 Apr 27. PMID 27132172

RESULTS

PARTICIPANT FLOW:
Groups:
- MXB Then PEG IFN: Myrcludex B 2mg daily for 24 weeks, followed by PEG IFN alfa-2a 180 µg/0.5 mL once weekly for 48 weeks
- MXB + PEG IFN Then PEG IFN: Myrcludex B 2mg daily and PEG IFN alfa-2a 180 µg/0.5 mL once weekly for 24 weeks, followed by PEG IFN alfa-2a 180 µg/0.5 mL once weekly for 24 weeks
Period: Overall Study
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Started | 8 | 8 | 8
Completed | 7 | 6 | 6
Not Completed | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.05) | 33.0 (4.87) | 42.1 (10.23) | 37.8 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 6
  Male | 5 | 7 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hepatitis B Surface Antigen (HBsAg) Response at Week 12 of Therapy
Description: HBsAg response was defined as serum HBsAg decline of at least 0.5 log IU/mL (or HBsAg negativation) at week 12 compared to baseline (including the patient with negative baseline level)
Time Frame: Baseline and 12 weeks
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Groups:
- MXB + PEG IFN Then PEG IFN: Myrcludex B 2mg daily and PEG IFN alfa-2a 180 µg/0.5 mL once weekly for 24 weeks, followed by pegINF 180mcg once weekly for 24 weeks
- PEG IFN: PEG IFN alfa-2a, 180 µg/0.5 mL once weekly for 48 weeks
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Hepatitis B Surface Antigen (HBsAg) Response at Week 24 of Therapy
Description: HBsAg response was defined as serum HBsAg decline of at least 0.5 log IU/mL (or HBsAg negativation) at week 24 compared to baseline (including the patient with negative baseline level)
Time Frame: Baseline and 24 weeks
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 8 | 8 | 8
Participants | 2 | 1 | 3

3. Secondary Outcome: Number of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) Response at Week 24 of Therapy
Description: HBV DNA response was defined as persistent reduction of HBV DNA by > 1 log IU/mL or negativation (including the patient with negative baseline level)
Time Frame: Baseline and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 8 | 8 | 8
Participants | 2 | 6 | 3

4. Secondary Outcome: Number of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) Response at Week 12 of Therapy
Description: as for outcome 3
Time Frame: Baseline and 12 weeks
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 8 | 8 | 8
Participants | 1 | 5 | 1

5. Secondary Outcome: Number of Participants With Hepatitis D Virus Ribonucleic Acid (HDV RNA) Response at Week 12 of Therapy
Description: HDV RNA response was defined as persistent reduction of HDV RNA by > 1 log IU/mL or negativation (including the patient with negative baseline level)
Time Frame: Baseline and 12 weeks
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 8 | 8 | 8
Participants | 4 | 5 | 6

6. Secondary Outcome: Number of Participants With Hepatitis D Virus Ribonucleic Acid (HDV RNA) Response at Week 24 of Therapy
Description: as for outcome 5
Time Frame: Baseline and 24 weeks
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 8 | 8 | 8
Participants | 7 | 7 | 7

7. Secondary Outcome: Number of Participants With Biochemical Response at Week 12 of Therapy
Description: Biochemical response was defined as normalization of ALT level as compared to baseline.
Time Frame: Baseline and 12 weeks
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 8 | 8 | 8
Participants | 2 | 2 | 2

8. Secondary Outcome: Number of Participants With Biochemical Response at Week 24 of Therapy
Description: Biochemical response was defined as normalization of ALT level as compared to baseline.
Time Frame: Baseline and 24 weeks
Population: For the efficacy assessments the main analysis set was Full analysis set (FAS): All patients of the Safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 8 | 8 | 8
Participants | 6 | 1 | 1

9. Secondary Outcome: Number of Participants With Covalently Closed Circular Deoxyribonucleic Acid (cccDNA) Response at Week 72 of Therapy
Description: Virological cccDNA response was defined as reduction of intrahepatic cccDNA by 0.5 log in comparison to baseline at the end of follow up.
Time Frame: Baseline and 72 weeks for arm A and 48 weeks for arms B and C
Population: No data to be reported due to absence of biopsy data. Biopsy data are unavailable because analyses were not performed
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | MXB Then PEG IFN | MXB + PEG IFN Then PEG IFN | PEG IFN
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MXB Then PEG IFN (N=8) | MXB + PEG IFN Then PEG IFN (N=8) | PEG IFN (N=8)
Leucopenia (Blood and lymphatic system disorders) | 7 (16) | 7 (11) | 7 (17)
Neutropenia (Blood and lymphatic system disorders) | 7 (17) | 7 (15) | 7 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (21) | 5 (14) | 6 (20)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (11) | 3 (4) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 3 (5) | 3 (4)
Gama-glutamyltransferase increased (Investigations) | 1 (1) | 2 (3) | 2 (5)
APTT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 5 (5) | 2 (2) | 3 (3)
Fatigue (General disorders) | 2 (2) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes